CLINICAL TRIAL: NCT03977532
Title: Study of a Red Blood Cell Deformability Parameter in Patients With Sickle Cell Disease, at Basal State and During Vaso-occlusive Crisis
Brief Title: Study of a Red Blood Cell Deformability Parameter in Patients With Sickle Cell Disease
Acronym: Drepaforme
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2018-36
Record Dates: First submitted 2019-06-03; First posted 2019-06-06 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with sickle cell disease (Experimental)
  Interventions: Other: Micro-blood sampling

INTERVENTIONS:
Other: Micro-blood sampling — capillary sampling of 40 microliters performed at the fingertip

SUMMARY:
Sickle cell disease is the most common genetic disease in the world. It results in the synthesis of an abnormal hemoglobin (HbS) which, in its deoxygenated form, polymerizes and causes structural changes in red blood cells (RBCs). They become more rigid and less deformable. The fragility of sickle-cell RBCs leads to their massive destruction, leading to chronic anemia (i.e. low hemoglobin in the blood) and to low tissue oxygenation. More rigid and less deformable, sickle-shaped RBCs tend to obstruct microvessels, leading to particularly painful vaso-occlusive crisis (VOC), which can cause organ failure (spleen, kidneys, brain, lungs, heart, liver, bone ...) and patient's lifethreatning. A preliminary work on red blood cells of sickle cell patients showed alteration of a parameter measuring the overall deformability of RBCs by assessing the nature of their movement in a shear flow. This parameter is altered sickle cell patients at basal state compared to a population of healthy individuals. This alteration is increased when sickle cell patients are in crisis.

The main objective of this project is to study the evolution of this parameter in sickle cell patients according to their health status (basal state vs vaso-occlusive crisis). The investigators hypothesize that the alteration of the RBC deformability parameter is significant before symptoms of vaso-occlusive crisis (several hours to several days). The main objective is a weekly analysis of the evolution of the parameter in 30 sickle cell patients (SS or SB°) in the basal state and daily in at least 6 patients at the beginning, during and just after a vaso-occlusive crisis. The comparison between the parameter measured in a subject in the basal state and in the same subject in crisis will be performed. The criteria for the presence of a vaso-occlusive crisis were: the appearance of a attacks of pain affecting at least two territories +/- fever> 38.3 +/- dyspnea and / or sputum. The investigators will differentiate the moderate VOC managed at home with low-level analgesics and VOC requiring hospitalization. The number of days of hospitalization, the occurrence of thrombotic complications, the degree of anemia and hemolysis will be noted. The measurement of the parameter will be performed on a capillary sampling of 40 microliters performed at the fingertip, weekly outside crises and daily when a crisis occurs.

ELIGIBILITY:
Inclusion Criteria:

* Homozygous SS or SB° sickle cell patients
* Person without regular blood transfusion

Exclusion Criteria:

* Other general diseases
* Psychiatric disorder
* Alcoholics
* Minors
* Absence of informed consent
* Pregnant or lactating woman
* Person under guardianship
* Person living in a health or social institution
* Person in emergency
* Person out of healthcare system
* Person deprived of liberty
* Person who has received a blood transfusion in the previous 3 months
* Person with regular blood transfusion or in a blood transfusion program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2023-08-03 (Actual)

PRIMARY OUTCOMES:
cytoplasmic viscosity measurement of red blood cells | 6 months
  Determination of the cytoplasmic viscosity parameter variations by measuring percentage of tanktreading (nature of movement of cells in a shear flow) from a micro-blood sample

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Garrido Pradalié, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France